CLINICAL TRIAL: NCT04975529
Title: Game on Philly: Engaging Underserved Middle School Youth in Out-of- School Time Sports and Nutrition Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 26406
Record Dates: First submitted 2021-06-03; First posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Exercise; Diet
MeSH Terms: conditions — Motor Activity | interventions — Nutrition Assessment

STUDY DESIGN:
Intervention Model Description: Two-group quasi-experimental
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Participants in intervention schools received access to daily, online after school programming, including live sessions with sports providers (via Zoom; rotating to provide exposure to multiple sports over the course of the intervention), weekly team meetings with a health coach (via Zoom), text-messages via the Remind app, and monthly delivery of Activity Kits with sports equipment, activity books, fresh produce, and incentives directly to their homes over 6-months.
  Interventions: Behavioral: Game on Philly: Engaging Underserved Middle School Youth in Out-of- School Time Sports and Nutrition Education
- Comparison Arm (Experimental): Participants in comparison schools received access to the Game on Philly app with workout and sports content that could be used asynchronously, and received one activity kit delivery with sports equipment and a self-guided activity book at the start of the program.
  Interventions: Behavioral: Game on Philly: Engaging Underserved Middle School Youth in Out-of- School Time Sports and Nutrition Education

INTERVENTIONS:
Behavioral: Game on Philly: Engaging Underserved Middle School Youth in Out-of- School Time Sports and Nutrition Education — Two-group quasi experimental intervention with schools assigned to intervention or comparison.

SUMMARY:
Game on Philly is a multi-component out-of-school time intervention delivered by trained sport-based youth development coaches and health navigators using evidenced-based programming. The program evaluation assesses the impact of this minimal-risk intervention to reduce the prevalence of obesity-related health disparities in racial and ethnic minority middle school youth. The program is a virtual sport-based youth development program, supplemented with nutrition education. The program was modified due to Covid-19 and is entirely virtual. Using a quasi-experimental design, six schools are assigned to the intervention arm and six schools are assigned to the comparison arm. Participants in intervention schools receive access to daily, online after school programming, with live sessions with sports providers (via Zoom), weekly team meetings with a health coach (via Zoom), text-messages via the Remind app, and the monthly delivery of Activity Kits directly to their homes for six months. Comparison school participants receive access to the Game on Philly app with workout and sports content and receive one activity kit delivery at the start of the program. Parent-child dyads recruited from each school complete surveys at baseline and at the end of the 6-month program (follow-up). It is hypothesized that youth participating in the intervention will experience significantly greater increases in physical activity at the end of the 6-month intervention compared to youth participating in the comparison arm (primary outcome). Secondary outcomes will examine changes in dietary intake, self-efficacy for physical activity and positive youth development.

ELIGIBILITY:
Inclusion Criteria (Parents) :

* 18 years of age or older
* Parent or legal guardian of the enrolled child
* Can read, write and speak in English

Inclusion Criteria (Child):

* Interested in and able to participate in the program for 6-months
* Can read, write and speak in English
* Are in 6th, 7th or 8th grade at a participating school

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2020-11-06 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in youth self-reported physical activity using the Patient-Reported Outcomes Measurement Information System (PROMIS) measure at 6-months | Change from baseline to end of the 6-month intervention
  Youth self-reported physical activity

SECONDARY OUTCOMES:
Mean change from baseline in youth self-reported self-efficacy for physical activity using the validated Physical Activity Self-efficacy scale at 6-months | Change from baseline to end of the 6-month intervention
  Youth self-reported self-efficacy for physical activity
Mean change from baseline in youth self-reported dietary intake assessed using the National Cancer Institute (NCI) fruit and vegetable screener at 6-months | Change from baseline to end of the 6-month intervention
  Youth self-reported dietary intake
Mean change from baseline in youth self-confidence assessed using the Positive Youth Development (PYD) Short Form Confidence scale at 6-months | Change from baseline to end of the 6-month intervention
  Youth self-reported confidence

CONTACTS AND LOCATIONS:
Overall Officials: Gina L Tripicchio, PhD, MSEd, Principal Investigator — Temple University
Locations (1):
- Temple University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No